CLINICAL TRIAL: NCT01784939
Title: HEPFER-Evaluation of a New Phenotypic Biological Marker in Genetic Type 1 Hemochromatosis
Acronym: HEPFER
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A01170-43
Record Dates: First submitted 2013-01-22; First posted 2013-02-06 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Hereditary Hemochromatosis C282Y Homozygous
Keywords: hereditary hemochromatosis C282Y homozygous; Iron Reabsorption Index (IRI); Hepcidin / ferritin (H / F) ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hepcidin serum ferritin serum transferrin serum iron serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HEPFER cohort: male, aged 18 and over, hereditary hemochromatosis C282Y homozygous diagnosed and followed in the service of Liver Diseases, University Hospital of Rennes
  - Maintenance therapy with phlebotomy for at least 1 year with stable iron stock on the basis of at least four previous plasma ferritin < 50μg / L

SUMMARY:
HFE(High iron FE)-related hereditary hemochromatosis has a highly variable penetrance. No phenotypic or genetic markers can predict the disease. The Iron Reabsorption Index (IRI), recently described by our group, correspond to the daily reabsorbed iron for a subject whose iron stock is stable and less than 50 µg / L.

The IRI is constant over time, reflecting the importance of the underlying functional deficit.

Hepcidin / ferritin (H / F) ratio may be an independent and constant over time marker of disease stage.No data are available on the validated values of this ratio.

The goal of this project is to determine the intra-individual variations of the H / F ratio over time during maintenance therapy and to assess the correlation with the IRI.

DETAILED DESCRIPTION:
HFE-related hereditary hemochromatosis has a highly variable penetrance : 1% of homozygous women and 30% of homozygous men would develop a clinically expressed disease. No predictive phenotypic or genetic markers are available.

The Iron Reabsorption Index (IRI), recently described by our group, correspond to the daily amount of reabsorbed iron for a subject whose iron stock is less than 50 µg / L and stabilized with maintenance phlebotomy.

For one patient, the IRI is constant over time, probably related to the functional deficit underlying. Unfortunately, IRI is a retrospective marker requiring at least one year of treatment, which limits its practical interest and directs its use for research activity.

We're looking for a more simple phenotypic marker readily available in clinical practice, which would predict at the time of diagnosis the evolution of the disease and therefore would better define the therapeutic options.

The pathophysiology of hemochromatosis is a dysregulation of hepcidin synthesis. We assume that hepcidin / ferritin ratio could be a phenotypic marker like the IRI, stage disease independent and constant over time. Indeed H/F ratio may reflect the adaptability of hepcidin production regulation for a level of iron stock No data are available on the validated values of this ratio. The aim of the project is to determine the intra-individual variations of the H / F ratio over time during maintenance therapy and to assess the correlation with the IRI.

The study involve 30 C282Y homozygous men, followed in a reference center with phlebotomy maintenance therapy and stabilized at a low level of ferritin (<50 µg / L) for at least 1 year.

The intra-individual variation of H/F ration will be determine by 5 samples every 14 days for 8 weeks. The correlation with IRI will be validated externally by the iron load observed at diagnosis. We will take into account other known variation factors like liver damages associated with hemochromatosis at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Men, at least 18 years old
* hereditary hemochromatosis C282Y homozygous diagnosed and followed in the service of Liver Diseases, University Hospital of Rennes
* Maintenance therapy with phlebotomy for at least 1 year with stable iron stock on the basis of at least four previous plasma ferritin < 50μg / L,
* Written, free and informed consent

Exclusion Criteria:

* Intercurrent illness unrelated to hemochromatosis causing cytolysis or inflammatory reaction.
* Person with a measure of legal protection (guardianship)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Men, at least 18 years old
  * hereditary hemochrmatosis C282Y homozygous diagnosed and followed in the service of Liver Diseases, University Hospital of Rennes
  * Maintenance therapy with phlebotomy for at least 1 year with stable iron stock on the basis of at least four previous plasma ferritin < 50μg / L,
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
distribution of values of Hepcidin / ferritin plasma ratio | First dosage on an empty stomach at current time of phlebotomy (Day 0), second dosage at day 14 at the same time, third dosage at day 28 at the same time, fourth dosage at day 42 at the same time, fifth dosage at day 56 at the same time
  values of Hepcidin / ferritin plasma ratio

SECONDARY OUTCOMES:
Correlation between Hepcidin / ferritin plasma ratio and IRI. | First dosage on an empty stomach at current time of phlebotomy (Day 0), second dosage at day 14 at the same time, third dosage at day 28 at the same time, fourth dosage at day 42 at the same time, fifth dosage at day 56 at the same time
Correlation between Hepcidin / Ferritin ratio before and after treatment | First dosage on an empty stomach at current time of phlebotomy (Day 0), second dosage at day 14 at the same time, third dosage at day 28 at the same time, fourth dosage at day 42 at the same time, fifth dosage at day 56 at the same time
Distribution of inter-individual Hepcidin / Ferritin ratio according to the stage of liver fibrosis | First dosage on an empty stomach at current time of phlebotomy (Day 0), second dosage at day 14 at the same time, third dosage at day 28 at the same time, fourth dosage at day 42 at the same time, fifth dosage at day 56 at the same time

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Jezequel, MD, Principal Investigator — CHU Rennes Pontchaillou
Locations (1):
- CHU, Rennes, France